CLINICAL TRIAL: NCT05968885
Title: Evaluation of the Efficacy and Urodynamic Outcomes Between Intradetrusor onabotulinumtoxinA Injection and Combination Pharmacotherapy in Patients With Detrusor Overactivity
Brief Title: Evaluation the Efficacy Between Botox Injection and Combination Pharmacotherapy in Patients With Detrusor Overactivity
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hui-Hsuan Lau, MD, Head of urogynecology, Associate Professor, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22MMHIS039e
Record Dates: First submitted 2023-03-02; First posted 2023-08-01 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2024-12

CONDITIONS: Urinary Bladder, Overactive; Urodynamics; Effect of Drug
Keywords: Detrusor overactivity; Urodynamic study; Combined pharmacotherapy; Botulinum Toxins; Effectiveness
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A; Injections; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intradetrusor onabotulinumtoxinA injection (Active Comparator): The toxin produced by Clostridium botulinum binds to the nerves endings and inhibits the muscular contractions, help to treat overactivity of the bladder muscles.
  Interventions: Procedure: Intradetrusor Botox® (onabotulinumtoxinA) injection
- Combination pharmacotherapy (Experimental): Combine Mirabegron and Solifenacin.
  Interventions: Drug: Combine Mirabegron and Solifenacin.

INTERVENTIONS:
Procedure: Intradetrusor Botox® (onabotulinumtoxinA) injection — The toxin produced by Clostridium botulinum binds to the nerves endings and inhibits the muscular contractions, help to treat overactivity of the bladder muscles.
  Arms: Intradetrusor onabotulinumtoxinA injection
Drug: Combine Mirabegron and Solifenacin. — Combination pharmacotherapy
  Arms: Combination pharmacotherapy

SUMMARY:
To investigates the effects of botulinum toxin type A bladder injection compared to combined pharmacotherapy with Mirabegron and Solifenacin.

DETAILED DESCRIPTION:
Patients with detrusor overactivity who were refractory to monotherapy with either anti-muscarinics or β3-adrenoceptor agonists were enrolled for prospective study. Patient were divided in two groups, intradetrusor onabotulinumtoxinA injection and combined pharmacotherapy with Mirabegron and Solifenacin. Incontinence-related symptoms distress and impact on quality of life were evaluated by short form of Urinary Distress Inventory, (UDI-6), Incontinence Impact Questionnaire (IIQ-7) and Overactive Bladder Symptom Score (OABSS). Objective outcomes include changes from baseline in daily urgency episodes, urinary incontinence episodes, maximum cystometric capacity, maximum detrusor pressure (Pdetmax) at first involuntary detrusor contraction and volume at first involuntary detrusor contraction were measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with detrusor overactivity which defined as a urodynamic observation characterized by involuntary detrusor contractions during the filling phase. Those who were refractory to monotherapy with either anti-muscarinics or β3-adrenoceptor agonists were enrolled for prospective study

Exclusion Criteria:

* Postvoid urine retention before treatment

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study focus on female detrusor overactivity.
Enrollment: 300 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Short form of Urinary Distress Inventory (UDI-6) | Assess before treatment and 1 month, 3 months, 6 months and 1 year after treatment
  UDI-6 is a valid questionnaire, used particularly to investigate symptoms associated with lower urinary tract dysfunction and inquire on irritative, stress, and obstructive or discomfort complaints. UDI-6 consists of six items: frequent urination; leakage related to feeling of urgency; leakage related to activity, coughing, or sneezing; small amounts of leakage (drops); difficulty emptying the bladder; and pain or discomfort in the lower abdominal or genital area. The total score ranges from 0 to 18 , with a higher score indicating more severe of incontinence.
Short form of Incontinence Impact Questionnaire (IIQ-7) | Assess before treatment and 1 month, 3 months, 6 months and 1 year after treatment
  The IIQ-7 assess the impact of urinary incontinence on QoL. 7 items assess influence of urinary incontinence on physical activity, travel, social/relationships & emotional health. Each item is scored between 0 (activities not affected at all) to 3 (activities greatly affected). The total score ranges from 0 to 21, with a higher score indicating more severe of incontinence.
Overactive Bladder Symptom Score (OABSS) | Assess before treatment and 1 month, 3 months, 6 months and 1 year after treatment
  The total OABSS is the sum of four symptom scores: daytime frequency (score 0-2), nighttime frequency (score 0-3), urgency (score 0-5), and urgency incontinence (score 0-5). The total score ranges from 0 to 15, with a higher score indicating more severe of OAB symptoms.

SECONDARY OUTCOMES:
Maximum cystometric capacity | Assess during 3 months - 1year after treatment
  One of the urodynamic measurement commonly used for describing the severity of detrusor overactivity
Maximum detrusor pressure at first involuntary detrusor contraction | Assess during 3 months - 1year after treatment
  One of the urodynamic measurement commonly used for describing the severity of detrusor overactivity
Volume at first involuntary detrusor contraction | Assess during 3 months - 1year after treatment
  One of the urodynamic measurement commonly used for describing the severity of detrusor overactivity

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Hsuan Lau, MD, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lightner DJ, Gomelsky A, Souter L, Vasavada SP. Diagnosis and Treatment of Overactive Bladder (Non-Neurogenic) in Adults: AUA/SUFU Guideline Amendment 2019. J Urol. 2019 Sep;202(3):558-563. doi: 10.1097/JU.0000000000000309. Epub 2019 Aug 8. PMID 31039103
- [Background] Mueller ER, van Maanen R, Chapple C, Abrams P, Herschorn S, Robinson D, Stoelzel M, Yoon SJ, Al-Shukri S, Rechberger T, Gratzke C. Long-term treatment of older patients with overactive bladder using a combination of mirabegron and solifenacin: a prespecified analysis from the randomized, phase III SYNERGY II study. Neurourol Urodyn. 2019 Feb;38(2):779-792. doi: 10.1002/nau.23919. Epub 2019 Jan 15. PMID 30644570
- [Derived] Hsieh MH, Hwang JC, Su TH, Lau HH. The Efficacy and Safety Between Intradetrusor OnabotulinumtoxinA Injection and Combined Pharmacotherapy in Patients With Refractory Overactive Bladder: A Randomized Controlled Trial. J Urol. 2025 Oct;214(4):344-353. doi: 10.1097/JU.0000000000004660. Epub 2025 Jul 1. PMID 40590342